CLINICAL TRIAL: NCT00249132
Title: Risperidone Versus Haloperidol Versus Placebo in the Treatment of Chronic Schizophrenia
Brief Title: A Study of the Effectiveness and Safety of Risperidone Compared With Haloperidol and Placebo in Patients With Chronic Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006067
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: chronic schizophrenia; psychotic disorder; risperidone; antipsychotic agents
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of different doses of risperidone (an antipsychotic medication) compared with placebo and with a fixed 20 mg/day dose of a standard antipsychotic, haloperidol, in patients with chronic schizophrenia.

DETAILED DESCRIPTION:
Chronic schizophrenia is a longer-term condition that is characterized by a lack of drive, underactivity and slowness, and social withdrawal. As with the acute form of schizophrenia, delusions and hallucinations are common. This is a randomized, double-blind, parallel-group study to evaluate the effectiveness and safety of four dosages of risperidone (2, 6, 10 or 16 mg/day) compared with placebo and with a fixed 20 mg/day dose of a standard antipsychotic, haloperidol in patients with chronic schizophrenia who are in-patients at the beginning of the study.

The study is composed of two phases: a 1-week period, in which patients receive placebo and all current medication for schizophrenia treatment is stopped, followed by a double-blind treatment phase. The doses of study drug are increased progressively during the first week of the double-blind period and then remain constant for the next 7 weeks. The primary measures of effectiveness are the percentage of patients showing clinical improvement (reduction of >=20% from baseline) on the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) and the total PANSS score, from baseline to end of double-blind treatment. The PANSS is a rating scale that measures the symptoms of schizophrenia. Safety evaluations include the incidence of adverse events, results of clinical laboratory tests (hematology, biochemistry, and urinalysis), plasma levels of risperidone, measurements of vital signs and body weight, physical examination and electrocardiogram (ECG) findings, neurological examinations, and the Extrapyramidal Symptoms Rating Scale (ESRS), a scale used to measure effects of antipsychotic medications on motor functions of the patient. The study hypothesis is that risperidone is more effective than placebo, as measured by clinical improvement on PANSS and the average total score for PANSS, in patients with chronic schizophrenia. Risperidone tablets, taken orally, starting with 1 mg twice daily, gradually increasing dose in Week 1 (except for 1 mg twice daily group), then 1, 3, 5, or 8 mg twice daily, continuing for 7 weeks. Haloperidol tablets, starting 1 mg twice daily and increasing to 10 mg twice daily (Week 1), continuing 10 mg twice daily for 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of chronic schizophrenic disorder, according to the Diagnostic and Statistical Manual of Mental Diseases, 3rd edition (DSM-III-R) criteria and are inpatients at the beginning of study
* total score on the PANSS (Positive and Negative Syndrome Scale for Schizophrenia) rating scale at study entry of >=60 and <=120
* females of childbearing age must demonstrate adequate birth control measures and have a negative pregnancy test before study entry.

Exclusion Criteria:

* Patients with mental disorders other than chronic schizophrenic disorder
* patients with clinically significant organic or neurological diseases
* patients with epilepsy
* history of alcohol or drug abuse history within the 6 months before study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Study Completion 1991-07 (Actual)

PRIMARY OUTCOMES:
Percent of patients showing clinical improvement, defined as a >=20% reduction in the total PANSS score from baseline to end of double-blind treatment, and the mean change from baseline to end of double-blind treatment in total PANSS score.

SECONDARY OUTCOMES:
Mean PANSS Positive Subscale Score; Mean PANSS Negative Subscale Score; mean PANSS General Psychopathology Subscale Score; CGI severity; CGI overall change from baseline; safety evaluations conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- [Result] Marder SR, Meibach RC. Risperidone in the treatment of schizophrenia. Am J Psychiatry. 1994 Jun;151(6):825-35. doi: 10.1176/ajp.151.6.825. PMID 7514366
- [Result] Chouinard G, Jones B, Remington G, Bloom D, Addington D, MacEwan GW, Labelle A, Beauclair L, Arnott W. A Canadian multicenter placebo-controlled study of fixed doses of risperidone and haloperidol in the treatment of chronic schizophrenic patients. J Clin Psychopharmacol. 1993 Feb;13(1):25-40. PMID 7683702
- [Result] Marder SR, Davis JM, Chouinard G. The effects of risperidone on the five dimensions of schizophrenia derived by factor analysis: combined results of the North American trials. J Clin Psychiatry. 1997 Dec;58(12):538-46. doi: 10.4088/jcp.v58n1205. PMID 9448657